CLINICAL TRIAL: NCT02248844
Title: Safety and Effectiveness of BOTOX® for Lateral Canthal Lines With or Without Simultaneous Glabellar Lines in Korea
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 191622-147
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Lateral Canthal Lines; Crow's Feet Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Botulinum Toxin Type A: Subjects who receive botulinum toxin Type A injected into crow's feet line areas per clinical practice.
  Interventions: Biological: Botulinum Toxin Type A

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Botulinum toxin Type A injected into crow's feet line areas per clinical practice.
  Other Names: BOTOX®; onabotulinumtoxinA

SUMMARY:
This is a postmarketing surveillance study in Korea to evaluate the safety and effectiveness of BOTOX® for lateral canthal lines (crow's feet lines) with or without simultaneous glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Subject and Investigator decision to treat crow's feet lines with Botox®

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Lateral Canthal Lines (Crow's Feet Lines)
Sampling Method: Non-Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2014-09-26 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 3 months

SECONDARY OUTCOMES:
Investigator's Assessment of Change in Appearance of Crow's Feet Lines on a 3-Point Scale | Baseline, Up to 3 months
Subject's Assessment of Change in Appearance of Crow's Feet Lines on a 7-Point Scale | Baseline, Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Dr. Robbin Clinic, Gangnam-gu, Seoul, South Korea

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com